CLINICAL TRIAL: NCT02222584
Title: The Effects of Physical Activity on Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0364
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2018-12

CONDITIONS: Inflammatory Bowel Disease
Keywords: inflammatory bowel disease; physical activity; disease activity; quality of life
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD group: patients with with inflammatory bowel disease who are visiting the out-patient clinic of severance hospital from July 2014 to February 2015

SUMMARY:
Physical activity (PA) is beneficial in the prevention and management of chronic disease. However, few data exist regarding the level of PA in inflammatory bowel disease (IBD) and whether or not vigorous PA may have beneficial effects on patients' health. To evaluate the level of PA and the effect of PA on disease activity of patients with IBD. To evaluate the effect of PA on quality of life of patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19
* patients with inflammatory bowel disease (Crohn's disease, Ulcerative Colitis, intestinal behcet's disease)

Exclusion Criteria:

* Age <19
* Patient who denied to response the survey questions
* Patient who denied to enroll the survey research

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with inflammatory bowel disease who are visiting the out-patient clinic of severance hospital from July 2014 to Feburary 2015
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2014-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
level of physical activity (PA) | 1 hour
  Physical activity (PA) levels were assessed using the International PA Questionnaire. Based on self-reported frequency (day) and duration (hr) of physical activities, corresponding metabolic equivalent (MET-hr/wk) values were calculated to lowest PA, low PA, moderate PA and highest PA

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea